CLINICAL TRIAL: NCT01584999
Title: Effects on the Septic Patient's Microcirculation of the Transfusion of Three Different Types of Concentrated Red Blood Cells.
Brief Title: Effects on Septic Patient's Microcirculation of the Transfusion of Different Types of Concentrated RBCs.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Prot 210163
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Septic Patients
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fresh not-leukocyte-reduced RBCs (Active Comparator)
  Interventions: Biological: Blood transfusion
- Fresh RBCs leukocyte-reduced (Active Comparator)
  Interventions: Biological: Blood transfusion
- RBCs with storage longer than 15 days (Active Comparator)
  Interventions: Biological: Blood transfusion

INTERVENTIONS:
Biological: Blood transfusion — RBCs have been transfused in septic patient admitted in ICU

SUMMARY:
Aim of the study is to evaluate the effects, on microcirculation of septic patient, of three types of RBCs: 1- fresh standard RBCs (storage <10 days); 2-leukodepleted RBCs and 3-old standard RBCs (storage >15 days) respectively. Before and 1 hour after the transfusion, microcirculation is evaluated using Sidestream Dark Field Imaging (SDF) and Near InfraRed Spectroscopy (NIRS) with vascular occlusion test. We also monitor temperature, heart rate, mean blood pressure, hemochrome, blood gases, blood lactates and SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis, severe sepsis or septic shock who, according to clinical evaluation, need a hemotransfusion.

Exclusion Criteria:

* Patients under 18 years of age; Pregnancy; Coagulative disorders; Cardiogenic shock (Met<4;)Acute massive bleeding (>8 U)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Microcirculatory Flow Index (MFI) before and after blood transfusion. | One hour after the end of blood transfusion compared with before blood transfusion
  Microcirculatory Flow Index detected in vivo by side-dark field imaging at sublingual microcirculation. It represents the quality of blood flow at microcirculatory level. This study wants to verify any of the considered different types of blood transfused can improve MFI.

SECONDARY OUTCOMES:
Perfused Vessel Density (PVD) | One hour after the end of blood transfusion compared with before blood transfusion
  Perfused Vessel Density detected in vivo by side-dark field imaging at sublingual microcirculation. It represents the quantity of well perfused vessels at microcirculatory level. This study wants to verify any of the considered different types of blood transfused can improve PVD.
StO2 upslope | One hour after the end of blood transfusion compared with before blood transfusion
  StO2 upslope is measured with Near InfraRed Spectroscopy at the tenar muscle. It represents the velocity of the recovery of the tissue oxygen saturation after a short period of ischemia of the hand, the Vascular Occlusion Test.
Arterial Blood Lactate | One hour after the end of blood transfusion compared with before blood transfusion
Arterial pH | One hour after the end of blood transfusion compared with before blood transfusion
SOFA score | One hour after the end of blood transfusion compared with before blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- University ICU, AOU Ospedali Riuniti, Torrette Di Ancona, Ancona, Italy

REFERENCES:
- [Derived] Damiani E, Adrario E, Luchetti MM, Scorcella C, Carsetti A, Mininno N, Pierantozzi S, Principi T, Strovegli D, Bencivenga R, Gabrielli A, Romano R, Pelaia P, Ince C, Donati A. Plasma free hemoglobin and microcirculatory response to fresh or old blood transfusions in sepsis. PLoS One. 2015 May 1;10(5):e0122655. doi: 10.1371/journal.pone.0122655. eCollection 2015. PMID 25932999
- [Derived] Donati A, Damiani E, Luchetti M, Domizi R, Scorcella C, Carsetti A, Gabbanelli V, Carletti P, Bencivenga R, Vink H, Adrario E, Piagnerelli M, Gabrielli A, Pelaia P, Ince C. Microcirculatory effects of the transfusion of leukodepleted or non-leukodepleted red blood cells in patients with sepsis: a pilot study. Crit Care. 2014 Feb 17;18(1):R33. doi: 10.1186/cc13730. PMID 24528648